CLINICAL TRIAL: NCT03127267
Title: Phase 3 Study to Compare the Efficacy and Safety of Masitinib in Combination With Riluzole Versus Placebo in Combination With Riluzole in the Treatment of Patients Suffering From Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Efficacy and Safety of Masitinib Versus Placebo in the Treatment of ALS Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB19001
Record Dates: First submitted 2017-04-13; First posted 2017-04-25 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; Tyrosine kinase inhibitor; Lou Gehrig's disease; Charcot's disease; Motor Neuron disease; MND
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — masitinib; Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Masitinib (4.5) & Riluzole (Experimental): Participants receive masitinib (3.0 mg/kg/day), given orally twice daily, with a dose escalation to 4.5 mg/kg/day after 4 weeks of treatment. Each ascending dose titration is subjected to a safety control. Masitinib will be administered as an add-on to riluzole at 50 mg b.i.d
  Interventions: Drug: Riluzole; Drug: Masitinib (4.5)
- Masitinib (6.0) & Riluzole (Experimental): Participants receive masitinib (3.0 mg/kg/day), given orally twice daily, with a dose escalation to 4.5 mg/kg/day after 4 weeks of treatment, followed by dose escalation to 6.0 mg/kg/day after 4 weeks of treatment. Each ascending dose titration is subjected to a safety control. Masitinib will be administered as an add-on to riluzole at 50 mg b.i.d.
  Interventions: Drug: Masitinib (6.0); Drug: Riluzole
- Placebo & Riluzole (Placebo Comparator): Participants receive a matched dose placebo, given orally twice daily, in combination with riluzole at 50 mg b.i.d.
  Interventions: Drug: Riluzole; Drug: Placebo

INTERVENTIONS:
Drug: Masitinib (6.0) — Masitinib (titration to 6.0 mg/kg/day)
  Other Names: AB1010
  Arms: Masitinib (6.0) & Riluzole
Drug: Riluzole — Riluzole 50 mg tablet, treatment per os
  Other Names: Rilutek
Drug: Placebo — treatment per os
  Other Names: Placebo Oral Tablet
  Arms: Placebo & Riluzole
Drug: Masitinib (4.5) — Masitinib (titration to 4.5 mg/kg/day)
  Other Names: AB1010
  Arms: Masitinib (4.5) & Riluzole

SUMMARY:
The objective is to compare the efficacy and safety of masitinib in combination with riluzole versus matched placebo in combination with riluzole for the treatment of Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
Masitinib is a selective, oral tyrosine kinase inhibitor with neuroprotective capability demonstrated via numerous preclinical studies. Two of masitinib's main cellular targets are the mast cell and microglia cell. It is well-established that mast cells play a prominent role in neuroinflammatory processes. Microglia, resident immune cells of the central nervous system (CNS), also constitute an important source of neuroinflammatory mediators and may have fundamental roles in numerous neurodegenerative disorders. The development of masitinib in ALS is therefore based on the pharmacological action of masitinib in microglia cells and mast cells, thereby slowing microglial-related disease progression, reducing neuro-inflammation, and modulating the neuronal microenvironment in both central and peripheral nervous systems. This is a multicenter, double-blind, randomized, placebo-controlled, parallel-group (two ascending dose titrations of masitinib and matching placebo), comparative study of oral masitinib in the treatment of patients with amyotrophic lateral sclerosis (ALS).

ELIGIBILITY:
Main inclusion criteria include:

* Patients diagnosed with laboratory supported probable, clinically probable or definite ALS according to the World Federation of Neurology Revised El Escorial criteria
* Patient with a familial or sporadic ALS
* ALS disease duration from diagnosis no longer than 24 months at the screening visit
* Patient treated with a stable dose of riluzole (100 mg/day) for at least 12 weeks days prior to the baseline visit
* Patient with an ALSFRS-R score progression between onset of the disease and screening of > 0.3 per month, confirmed with an ALSFRS-R score progression of ≥ 1 point during a 12-week run-in period between screening and randomization.
* Patient with a score, at screening, of at least 26 overall, including a score of at least 3 on item #3 and at least 2 on each of the 12 ALSFRS-R individual component items and with a score, at randomization, of at least 2 on each of the 12 ALSFRS-R individual component items

Main exclusion criteria include:

* Patient with dementia or significant neurological, psychiatric, systemic or organic disease, uncontrolled or that may interfere with the conduct of the trial or its results
* Patient with a FVC < 60% predicted normal value for gender, height, and age at screening and baseline
* Pregnant, or nursing female patient

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
ALSFRS-R | 48 weeks
  Change in Amyotrophic Lateral Sclerosis functional rating scale (ALSFRS)-Revised.

SECONDARY OUTCOMES:
ALSAQ-40 | 48 weeks
  Change in ALS quality of life patient questionnaire (ALSAQ-40)
PFS | From day of randomization to disease progression or death, assessed for a maximum of 36 months
  Progression free survival (PFS) is defined as the time from randomization to progression (decline of more than 9 points in ALSFRS-R score from baseline) or death
FVC | 48 weeks
  Change in Forced Vital Capacity (FVC)
HHD | 48 weeks
  Change in evaluation of upper- and lower-limb muscle strength using hand-held dynamometry (HHD)
Change in the Combined Assessment of Function and Survival (CAFS) score from baseline to week 48 | 48 weeks
  CAFS ranks patients' clinical outcomes based on survival time and change in the ALS Functional Rating Scale-Revised (ALSFRS-R) score. Each patient's outcome is compared to every other patient's outcome, assigned a score, and the summed scores are ranked. The mean rank score for each treatment group can then be calculated. A higher mean CAFS score indicates a better group outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Ludolph, MD, PhD, Principal Investigator — Department of Neurology, University of Ulm, Germany
Locations (56):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Medicine Brain Science Institute, Baltimore, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Virginia Health System, Charlottesville, Virginia
- University Hospital Leuven (UZ Leuven), Leuven, Belgium
- Bispebjerg Hospital, Copenhagen, Denmark
- France (11):
  - CHU de Angers, Angers
  - Groupe Hospitalier Pellegrin Tripode, Bordeaux
  - Hôpital neurologique Pierre Wertheimer, Bron
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHU de Lille - Hopital Roger Salengro, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - CHU de Marseille - Hôpital de la Timone, Marseille
  - CHRU de Montpellier - Gui de Chauliac, Montpellier
  - CHU de Nancy - Hopital Central, Nancy
  - CHU Hôpital Pasteur Nice, Nice
  - CHRU de Tours - Hopital Bretonneau, Tours
- Department of Neurology, University of Ulm, Ulm, Germany
- Greece (4):
  - Athens Naval Hospital, Athens
  - Eginition Hospital, Athens
  - University General Hospital of Larissa, Larissa
  - General University Hospital of Patras, Rio
- Israel (2):
  - Hadassah University Hospital, Jerusalem
  - Tel-Aviv Medical Center Hôpital Sourasky (ICHILOV), Tel Aviv
- Italy (11):
  - Ospedale Civile Sant'Agostino - Estense, Baggiovara, Modena
  - ASST degli Spedali Civili di Brescia, Brescia
  - Centro Clinico NeMO Fondazione Serena Onlus, Gussago
  - Clinico Nemo Center (Centro Clinico NeMO Milano), Milan
  - IRCCS Istituto Auxologico Italiano, Milan
  - Istituti Clinici Scientifici Maugeri IRCCS, Milan
  - San Raffaele Hospital (Ospedale San Raffaele), Milan
  - University Hospital Maggiore della Carita, Novara
  - Azienda Ospedale-Università Padova, Padua
  - IRCCS Mondino Foundation, Pavia
  - University Hospital in Turin (Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino), Torino
- Oslo University Hospital HF Ullevål, Oslo, Norway
- Centrum Medyczne Neuromed, Bydgoszcz, Poland
- Hospital de Santa Maria, Lisbon, Portugal
- Russia (2):
  - Moscow city clinical Hospital after V.M. Buyanov, Moscow
  - Scientific Practical Medical Center "Innovation and Health", Novosibirsk
- Clinical Centre of Serbia, Belgrade, Serbia
- Klinicni center Ljubljana, Ljubljana, Slovenia
- Spain (6):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Carlos III, Madrid
  - Hospital San Rafael, Madrid
  - Clinical Hospital Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario y Politecnico La Fe, Valencia
- Sweden (3):
  - Centralsjukhuset Karlstad (Central Hospital Karlstad), Karlstad
  - Skåne University Hospital, Malmo
  - Norrlands universitetssjukhus, Umeå
- Ukraine (3):
  - The State Institution of Neurology, Psychiatry and Narcology of NAMS of Ukraine, Kharkiv
  - Medical Center of LLC Medical Center Dopomoga Plus, Kyiv
  - Communal Non-Profit Enterprise of Lviv Regional Council, Lviv Regional Clinical Hospital, Neurological Department, Lviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Latham BD, Oskin DS, Crouch RD, Vergne MJ, Jackson KD. Cytochromes P450 2C8 and 3A Catalyze the Metabolic Activation of the Tyrosine Kinase Inhibitor Masitinib. Chem Res Toxicol. 2022 Sep 19;35(9):1467-1481. doi: 10.1021/acs.chemrestox.2c00057. Epub 2022 Sep 1. PMID 36048877